CLINICAL TRIAL: NCT04809701
Title: Evaluation of Different Defibrillation Electrode Configurations for Development of a Non-vascular ICD
Brief Title: Non-vascular ICD Electrode Configuration Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10369
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Ventricular Arrythmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Configuration A first (Experimental): Subjects receive the test of Configuration A first and Configuration B second.
  Interventions: Procedure: Temporary implantation of defibrillation coils and pulse generator; Procedure: Defibrillation following induction of VA (Configuration A first); Procedure: Removal of defibrillation coils and pulse generator
- Configuration B first (Experimental): Subjects receive the test of Configuration B first and Configuration A second.
  Interventions: Procedure: Temporary implantation of defibrillation coils and pulse generator; Procedure: Defibrillation following induction of VA (Configuration B first); Procedure: Removal of defibrillation coils and pulse generator

INTERVENTIONS:
Procedure: Temporary implantation of defibrillation coils and pulse generator — Each subject will undergo temporary implantation of defibrillation coils and pulse generator according to the NV-ICD electrode configurations.
Procedure: Defibrillation following induction of VA (Configuration A first) — Ventricular arrhythmia (VA) will be induced via an EP catheter placed in the right ventricle. After VA is confirmed, a defibrillation shock will be attempted to terminate the arrhythmia. Up to two defibrillation energies will be tested for Configuration A. Then up to two defibrillation energies will be tested for Configuration B.
  Arms: Configuration A first
Procedure: Defibrillation following induction of VA (Configuration B first) — Ventricular arrhythmia (VA) will be induced via an EP catheter placed in the right ventricle. After VA is confirmed, a defibrillation shock will be attempted to terminate the arrhythmia. Up to two defibrillation energies will be tested for Configuration B. Then up to two defibrillation energies will be tested for Configuration A.
  Arms: Configuration B first
Procedure: Removal of defibrillation coils and pulse generator — Defibrillation coils and pulse generator will be removed from the subject after the defibrillation tests are completed.

SUMMARY:
This study is designed to evaluate the energy requirements of two different Nonvascular ICD (NV-ICD) electrode configurations for achieving successful defibrillation of ventricular arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. Patient that is scheduled to undergo surgery requiring midline sternotomy or implantation of a commercially-available TV-ICD or S-ICD system per local guidelines
2. Patient must be at least 18 years of age
3. Subject must provide written informed consent prior to any clinical investigation-related procedure.

Exclusion Criteria:

1. Pacemaker dependency
2. Chronically implanted cardiac implantable electronic device or other device which delivers an electrical current
3. Currently taking amiodarone or a Class IC antiarrhythmic drug
4. Hypertrophic cardiomyopathy
5. Anticipated high risk of stroke
6. Anticipated high surgical risk or risk of infection
7. Severe aortic stenosis
8. Severe proximal three vessel coronary disease (over 70% in each vessel)
9. Greater than 50% left main stem disease
10. Prior surgery or anatomical abnormality that significantly increases implant risk per physician's discretion
11. Medical conditions that preclude defibrillation testing
12. Chronic renal insufficiency including patients on dialysis
13. Subject is currently participating in another clinical investigation.
14. Pregnant or nursing subjects and those who plan pregnancy during the clinical investigation follow-up period.
15. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with the 1-month phone follow-up requirements of the clinical investigation results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
The rate of successful defibrillation of induced VA using each of the two NV-ICD electrode configurations | During the study procedure
  Successful defibrillation is defined as termination of the induced VA to sinus rhythm or other non-life threatening ventricular or escape rhythm (such as atrial fibrillation) as determined by the implanting physician.

OTHER OUTCOMES:
The number of acute adverse events associated with the temporary implant and defibrillation testing with the two NV-ICD electrode configurations under investigation | Within 1 month of the study procedure
  Descriptive outcome summarizing possible acute adverse events with the temporary implant and defibrillation testing

CONTACTS AND LOCATIONS:
Overall Officials: Reinoud E Knops, MD, PhD, Principal Investigator — Academic Medical Center Department of Cardiology Meibergdreef 9 1105 AZ Amsterdam The Netherlands
Locations (3):
- Hospital Clínico Regional de Concepción, Concepción, Bio Bio, Chile
- Na Homolce Hospital, Prague, Czechia
- Centro de Intervenciones Endovasculares y Cirugía Cardiovascular, Asunción, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No